CLINICAL TRIAL: NCT05725499
Title: Neuromodulation of Blood Pressure Using Transcutaneous Spinal Stimulation in Chronic Spinal Cord Injury
Brief Title: The Effect of Transcutaneous Stimulation on Blood Pressure in Spinal Cord Injury (SCI)
Acronym: SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Einat Haber, Associate Research Scientist, Kessler Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R.1197.22; PC8-23 (Other Grant/Funding Number: New Jersey Health Foundation)
Record Dates: First submitted 2023-01-25; First posted 2023-02-13 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries; Hypotension; Orthostatic Hypotension; Spinal Cord Diseases; Cardiovascular Diseases; Trauma, Nervous System; Central Nervous System Diseases; Nervous System Diseases; Blood Pressure
Keywords: Transcutaneous Spinal Cord Stimulation; Spinal Stimulation; Orthostatic Hypotension; Blood Pressure; Neuromodulation
MeSH Terms: conditions — Spinal Cord Injuries; Hypotension; Hypotension, Orthostatic; Spinal Cord Diseases; Cardiovascular Diseases; Trauma, Nervous System; Central Nervous System Diseases; Nervous System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with a chronic SCI (≥ 6 months after injury) (Experimental): Participants will complete three days of baseline assessments (including a baseline orthostatic test and a day of neurophysiological mapping), five days of stimulation mapping to locate the optimal spinal sites for a blood pressure response, a day of testing with stimulation applied during an orthostatic provocation and a two-week (total of six days) training period with repeated exposure to stimulation, followed by two days of additional orthostatic tests (with and without stimulation)
  Interventions: Device: Biostim-5 transcutaneous spinal stimulator; Diagnostic Test: Tilt-table orthostatic stress testing

INTERVENTIONS:
Device: Biostim-5 transcutaneous spinal stimulator — Transcutaneous stimulation of the spinal cord. Mapping will be performed to determine sites for optimal modulation of blood pressure. During each mapping day, with participants in a supine or seated position, electrodes will be placed on the midline of one of the following spinous processes: C5/6, T7/8, T11/12, L1/2 and S1/2. Stimulation intensity will start at 5 mA and gradually increased in 5 mA increments up to 100 mA. The frequency will be 2 or 30 Hz. Profiles will be established to guide selection of optimal site locations for blood pressure modulation. The profile chosen will be used during training and testing.
  During testing, stimulation will be applied using the selected profile in order to normalize SBP to the range of 110-120 mmHg and stabilize it within this range during a 30-min tilt test.
  On each session during the 2-week training-period, stimulation will be applied for 30 minutes using the selected profile, while the participant remains in a seated position.
Diagnostic Test: Tilt-table orthostatic stress testing — While lying supine, participants will be strapped to a Hi-Low tilt-table bed. The bed will gradually be tilted to a 70 degrees tilt, during which time continuous hemodynamic measures will be recorded. This position will be maintained for 30 minutes.
  During some of the sessions, the tilt test will be accompanied by spinal stimulation.

SUMMARY:
This project will investigate the effect of spinal cord transcutaneous stimulation on blood pressure in individuals with a chronic spinal cord injury who experience blood pressure instability, specifically, orthostatic hypotension (a drop in blood pressure when moving from lying flat on your back to an upright position).

The main questions it aims to answer are:

1. What are the various spinal sites and stimulation parameters that normalize and stabilize blood pressure during an orthostatic provocation (70 degrees tilt)?
2. Does training, i.e., exposure to repeated stimulation sessions, have an effect on blood pressure stability?

Participants will undergo orthostatic tests (lying on a table that starts out flat, then tilts upward up to 70 degrees), with and without stimulation, and changes in their blood pressure will be evaluated.

DETAILED DESCRIPTION:
Cardiovascular (CV) control in persons with a high level (thoracic level T6 or above) spinal cord injury (SCI) is often impaired, resulting in short and long-term health complications and a decline in quality of life. Orthostatic hypotension (OH), a significant decrease in blood pressure (BP) when moving from lying flat (supine) to an upright position, appears early after injury and is frequently accompanied by dizziness, weakness, fatigue, and even syncope. In the long term, while symptoms are typically diminished, it still clinically occurs in 50% of individuals with a cervical injury. The physical, social, and emotional consequences of OH pose a major issue. Moreover, BP instability is associated with a decline in CV health and somewhat accounts for the 3 to 4-fold increased risk for stroke and heart disease in this clinical population.

In recent years, epidural spinal cord stimulation has been explored with promising results as a potential treatment for CV dysfunction. Spinal cord transcutaneous stimulation (scTS) represents an alternate approach, with the potential to benefit more people with fewer risks. Only one study thus far successfully applied scTS to restore CV function and resolve orthostatic symptoms following SCI, with stimulation applied at one thoracic location.

The objective of this study is to investigate the effect of scTS on BP in individuals with chronic SCI who experience OH. Stimulation sites and parameters that consistently increase and stabilize systolic BP within the range of 110-120 mmHg, during an orthostatic provocation (a 70° tilt-test), will be sought. The investigators will also evaluate whether there is any change in the BP response following repeated stimulation sessions. This project will provide the foundational evidence to use scTS to improve autonomic function in various SCI populations and help overcome barriers to engagement in activity and participation imposed by autonomic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury for greater than or equal to 6 months
* Injury level ≥ T6 (thoracic level)
* American Spinal Injury Association (ASIA) Impairment Scale (AIS) A-D
* Exhibits at least one of the following hypotensive symptoms:

  1. Baseline hypotension - resting supine or seated systolic blood pressure(SBP) < 90mmHg;
  2. SBP drop ≥ 20 mmHg within 5 minutes of assuming seated position;
  3. Symptoms of orthostasis with a drop of SBP (<90mmHg) from supine to sitting

Exclusion Criteria:

* Current illness (infection, a pressure injury that might interfere with the intervention, a recent diagnosis of DVT/PE, etc.)
* Ventilator-dependent
* History of implanted brain/spine/nerve stimulators
* Cardiac pacemaker/defibrillator or intra-cardiac lines
* Significant coronary artery or cardiac conduction disease, a recent history of myocardial infarction
* Insufficient mental capacity to understand and independently provide consent
* Pregnancy
* Cancer
* Deemed unsuitable by study physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Optimal stimulation sites | Through Mapping and testing sessions, average of 3 weeks
  Identify scTS spinal segments that restore systolic BP within the normotensive range (110-120 mmHg).
Optimal stimulation frequency | Through Mapping and testing sessions, average of 3 weeks
  Identify scTS frequency that restores systolic BP within the normotensive range (110-120 mmHg).
Systolic blood pressure - efficacy of stimulation | Throughout the experiment, average of 6 weeks
  Evaluate changes in blood pressure during an orthostatic test (comparing measurements obtained during stimulation to those obtained without).
  The ability of scTS to normalize SBP (to the range of 110-120) and to stabilize it over the course of a 30-min tilt test will be assessed.
Systolic blood pressure - effect of training | Post training, average of 2 weeks
  Explore the blood pressure response to orthostatic stress with and without stimulation, following six days of repetitive 30-min customized scTS sessions
Orthostatic symptoms questionnaire | Throughout the experiment, average of 6 weeks
  A questionnaire ranking the severity of orthostatic symptoms (dizziness, nausea), with a scale of 1-10 (10 being the most severe).

SECONDARY OUTCOMES:
EMG of leg muscles - muscle activation (analysis of mean and peak amplitudes) | Through Mapping and testing sessions, average of 3 weeks
  Analysis of leg-muscle EMG to identify configurations that modulate BP without eliciting motor activity, to ensure that BP response was not due to lower limb muscle contraction.
Spinal Cord Injury-Quality of Life (SCI-QOL) questionnaires | Before the first session and after the last session, average of 6 weeks
  Accessible through computer adaptive testing and addresses the following domains: emotional health, physical-medical health, social participation, and physical function
Global response assessment (GRA) | post training, average of 6 weeks
  GRA will be used to evaluate patients' perceptions of treatment effectiveness
Additional hemodynamic measure - diastolic blood pressure | throughout the trial, average of 6 weeks
  Hemodynamic measures will be collected throughout the trial
Additional hemodynamic measure - heart rate | throughout the trial, average of 6 weeks
  Hemodynamic measures will be collected throughout the trial

CONTACTS AND LOCATIONS:
Overall Officials: Gail F Forrest, Phd, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No